CLINICAL TRIAL: NCT07329517
Title: Comparative Effects of Resistance Training and Neuromuscular Training on Power, Knee Function and Dynamic Balance in Runners With Patellofemoral Syndrome
Brief Title: Comparative Effects of Resistance Training and Neuromuscular Training in Runners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0494
Record Dates: First submitted 2025-12-29; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: resistance training; neuromuscular training; runners
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Randomized control design
Who Masked: Outcomes Assessor
Masking Description: The Outcome Assessors are blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): 19 participants will be in group 1 and allocated for resistance training group (RT Group)
  Interventions: Other: Resistance training
- Group B (Active Comparator): 19 participants will be in group B and allocated for neuromuscular training (NT Group)
  Interventions: Other: Neuromuscular Training

INTERVENTIONS:
Other: Resistance training — 19 participants will be in group A and allocated for resistance training
  Arms: Group A
Other: Neuromuscular Training — 19 participants will be in group B and allocated for neuromuscular training
  Arms: Group B

SUMMARY:
This randomized controlled trial will include a sample of 38 young runners, calculated using epitool. Participants will be recruited through non-probability convenient sampling and randomly assigned to one of two groups: Group A (runner-specific resistance training) and Group B (neuromuscular training), with 19 participants in each group. The study will be conducted at the University of Lahore.

DETAILED DESCRIPTION:
The objective of this study is to compare the effects of resistance training and neuromuscular training on Power, Knee function and dynamic balance in runners with patellofemoral pain syndrome This randomized clinical trial will include a sample of 38 young runners, calculated using epitool.

Participants will be recruited through non-probability convenient sampling and randomly assigned to one of two groups: Group A (runner-specific resistance training) and Group B (neuromuscular re-education training), with 19 participants in each group. The study will be conducted at the University of Lahore. Inclusion criteria include male and female runners aged 18-30 with at least one years of running experience and no serious injuries in the past six months. Exclusion criteria include current injuries, medical conditions, or involvement in conflicting training programs. Pre- and post-intervention assessments will include the vertical jump test, IKDC questionnaire and SEBT test .Both groups will train three times per week over six weeks, with sessions supervised by qualified coaches for safety and adherence. All participants will provide written informed consent, ensuring confidentiality. This research seeks to inform training strategies in runners, providing insights that may improve performance outcomes for young runners and guide trainers in selecting effective training methods. It also aims to raise awareness of the diverse benefits of different training approaches, potentially increasing youth participation in running and contributing to sports science literature on effective conditioning practices.

ELIGIBILITY:
Inclusion Criteria:

* Runners aged 18-30 years
* Runners having at least one year of playing
* Male Runners with Patellofemoral pain syndrome
* Not involved in resistance or neuromuscular training

Exclusion Criteria:

* Individuals with other acute or chronic knee injuries
* history of knee surgery
* Runners who have not been consistently running for at least 6 months prior to the study

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 38 (Actual)
Dates: Start 2024-11-21 (Actual); Primary Completion 2025-10-05 (Actual); Study Completion 2025-11-05 (Actual)

PRIMARY OUTCOMES:
vertical Jump Test | 6 weeks
  The vertical jump test measures explosive leg power by comparing an athlete's standing reach with the height they achieve when jumping. The difference between these two points indicates their vertical jump height, which reflects lower-body strength and is commonly used in sports to assess athletic performance potential.
IKDC questionnaire | 6 weeks
  The IKDC questionnaire is a patient-reported tool that measures knee symptoms, daily function, and sports activity, producing a score from 0 (severe problems) to 100 (optimal function). It is widely used in orthopedics to track recovery and compare treatment outcomes for various knee conditions.
Star excursion balance test (SEBT) | 6 weeks
  The Star Excursion Balance Test (SEBT) is a dynamic assessment of balance and lower-limb function. In the test, a person stands on one leg and reaches in multiple directions with the other leg, challenging stability, strength, and flexibility. It is commonly used in sports and rehabilitation to detect injury risks, evaluate postural control, and monitor recovery progress.

CONTACTS AND LOCATIONS:
Overall Officials: Haleema Najeeb, DPT, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - The University of Lahore, Lahore, Punjab Province
  - University of Lahore, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bolgla LA, Boling MC. An update for the conservative management of patellofemoral pain syndrome: a systematic review of the literature from 2000 to 2010. Int J Sports Phys Ther. 2011 Jun;6(2):112-25. PMID 21713229
- [Background] Coburn SL, Barton CJ, Filbay SR, Hart HF, Rathleff MS, Crossley KM. Quality of life in individuals with patellofemoral pain: A systematic review including meta-analysis. Phys Ther Sport. 2018 Sep;33:96-108. doi: 10.1016/j.ptsp.2018.06.006. Epub 2018 Jun 28. PMID 30059951
- [Background] Rabelo ND, Lima B, Reis AC, Bley AS, Yi LC, Fukuda TY, Costa LO, Lucareli PR. Neuromuscular training and muscle strengthening in patients with patellofemoral pain syndrome: a protocol of randomized controlled trial. BMC Musculoskelet Disord. 2014 May 16;15:157. doi: 10.1186/1471-2474-15-157. PMID 24884455
- [Background] Clijsen R, Fuchs J, Taeymans J. Effectiveness of exercise therapy in treatment of patients with patellofemoral pain syndrome: systematic review and meta-analysis. Phys Ther. 2014 Dec;94(12):1697-708. doi: 10.2522/ptj.20130310. Epub 2014 Jul 31. PMID 25082920
- [Background] Rixe JA, Glick JE, Brady J, Olympia RP. A review of the management of patellofemoral pain syndrome. Phys Sportsmed. 2013 Sep;41(3):19-28. doi: 10.3810/psm.2013.09.2023. PMID 24113699
- [Background] Luo Y, Chen X, Shen X, Chen L, Gong H. Effectiveness of Kinesio tape in the treatment of patients with patellofemoral pain syndrome: A systematic review and meta-analysis. Medicine (Baltimore). 2024 Jun 7;103(23):e38438. doi: 10.1097/MD.0000000000038438. PMID 38847704
- [Background] Masoudi A, Chemane N, Useh U, Bello B, Magida N. Effectiveness of Self-Management Programs Among Athletes With Patellofemoral Pain Syndrome: Protocol for a Systematic Review. JMIR Res Protoc. 2024 Nov 1;13:e58340. doi: 10.2196/58340. PMID 39485375
- [Background] Nunes GS, de Moraes WSLA, de Souza Sampaio V, Seda NR, Dos Santos Mouta G, Dangui AJM, de Souza Petersen R, Nakagawa TH. Are Changes in Dynamic Knee Movement Control Related to Changes in Pain or Function in People With Knee Disorders? A Systematic Review and Meta-analysis. J Orthop Sports Phys Ther. 2023 Jul;53(7):388-401. doi: 10.2519/jospt.2023.11628. PMID 37068162